CLINICAL TRIAL: NCT06791694
Title: Comparison of Color Measurements of Postgraduate Dental Students in the Maxillary Anterior Region Using Different Color Determination Methods
Brief Title: Comparison of Color Measurements of Postgraduate Dental Students Using Different Color Determination Methods
Acronym: Color
Status: Enrolling by invitation | Type: Observational
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Kemal Işıklı, Research Asisstant, Hacettepe University
Other Study IDs: KA-21049
Record Dates: First submitted 2025-01-19; First posted 2025-01-24 (Actual); Last update posted 2025-01-30 (Actual); Status verified 2025-01

CONDITIONS: Tooth Discoloration
Keywords: color; tooth; button
MeSH Terms: conditions — Tooth Discoloration | interventions — Composite Resins

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Resins, Composite — Graduate students; healthy maxillary central teeth and color measurements will be performed with 4 different methods in at least 32 patients aged between 18-40 years. Firstly, students will be asked to make color measurements using the traditional method with two different color scales (Vita classical and Vita 3D master). As the third method; the enamel color of the teeth will be determined on digital photographs using the buton technique. Finally, tooth color will be measured on the buccal surface of the central teeth using a spectrophotometer.
  Other Names: vita classical; Vita 3D master; spectrophotometer

SUMMARY:
This study evaluates the accuracy of tooth color identification skills in the anterior region using a new technique, the button technique, in comparison with other methods.

DETAILED DESCRIPTION:
The human eye is effective in detecting subtle differences in tooth color. However, variations in the shade, translucency, opacity, and characterization of a tooth may not be accurately identified. Visual color matching is subject to physiological variables that may lead to inconsistencies, such as age, gender, experience, the type of scale used, varying degrees of light exposure, eye fatigue, and color vision deficiency.

Studies comparing visual and instrumental methods have demonstrated that spectrophotometers yield better results compared to visual color scales. Therefore, it is expected that color measurement devices improve the accuracy of tooth color determination, thereby enhancing the interpretation and aesthetic execution of restorations.

In recent years, the button technique has been described for shade selection in direct aesthetic restorations in the anterior region. In this technique, small composite samples in the form of dots are polymerized on the tooth surface using a curing light. Digital photographs are then taken, and appropriate enamel and dentin shades are selected on a computer using polarized and black-and-white images.

Very few clinical studies have investigated the use of digital color images obtained through intraoral digital scanners for shade selection, comparing them with other existing methods.

The aim of this study is to evaluate the accuracy of shade determination skills in the anterior region by comparing a new technique, the button technique, with other methods and to recommend the most suitable method for shade selection

ELIGIBILITY:
Inclusion Criteria:

* Being healthy individuals,
* Not having any systemic diseases,
* Being young individuals (18-40 age range)
* Vital, decay-free and healthy upper central teeth,
* Absence of caries-free hard tissue abrasions, any restoration, fracture, crack, intrinsic or extrinsic discoloration in the upper central teeth
* Lack of removable prosthesis feet for central teeth

Exclusion Criteria:

* Tetracycline, fluorosis staining of upper central teeth
* Patients with dentin exposure or loss of bine in the upper central teeth for any reason
* Pregnant and lactating patients will not be included.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Being healthy individuals, not having any systemic diseases, being young individuals (18-40 age range)
Sampling Method: Probability Sample
Enrollment: 32 (Estimated)
Dates: Start 2025-01-27 (Actual); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
To have compared the inter-observer reliability of 4 different methods used in tooth color selection | 1 month
  To have compared the inter-observer reliability of 4 different methods used in tooth color selection

CONTACTS AND LOCATIONS:
Locations (1):
- Hacettepe University, Altındağ, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided